CLINICAL TRIAL: NCT01542359
Title: Effectiveness of Yoga on Ambulatory Blood Pressure in Patients With Pre- and Stage I Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Long Island University (Other)
Responsible Party: Principal Investigator, Marshall Hagins, Professor, Long Island University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1SC3GM088049-01A1 REVISED; 1SC3GM088049-01A1 (NIH)
Record Dates: First submitted 2012-02-19; First posted 2012-03-02 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension
Keywords: Yoga, Hypertension; Blood Pressure; Autonomic Nervous system
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): The integrated yoga program was designed to: 1) include the three primary elements of yoga as most commonly practiced in western cultures (physical postures, breath control and meditation); and 2) be appropriate for those without any prior yoga experience and with pre- and Stage I hypertension. The yoga program was designed by Eddie Stern, Founder and Director of "Ashtanga Yoga New York" (AYNY) in consultation with Drs. Hagins and Rundle, and are in large part congruent with the yoga program we studied previously (see Preliminary Studies). The yoga class includes: instruction on yogic principles regarding moral precepts (yamas and niyamas); active postures requiring mild-moderate physical exertion; conscious control of the breath in synchrony with active postures; and meditation. We expect approximately 10-15 minutes of the integrated yoga program to consist of isolated practice of meditation (occurring independently of the moving postures, typically in seated or lying positions).
  Interventions: Other: Yogic practice
- Conventional Exercise (Active Comparator): Conventional exercise such as standing toe touch with arm swings, curl ups, push ups, leg lifts, etc. All done at a relatively slow rate which will be non-aerobic and at an average rate across the session of 3 METs
  Interventions: Other: Conventional Exercise

INTERVENTIONS:
Other: Yogic practice — breathing, meditation, physical postures
  Arms: Yoga
Other: Conventional Exercise — Standard physical exercises such as toe touch in standing, curl ups, push ups, leg lifts
  Arms: Conventional Exercise

SUMMARY:
The proposed study will compare a well defined and integrated yoga practice (postures/breath control/meditation) to a conventional exercise program in reducing hypertension. The expected outcomes include data on the effects of yoga on ambulatory blood pressure, psychosocial stress, and the autonomic system in individuals with pre- and Stage I hypertension. The information gained in this study will have a positive impact by providing critical preliminary and feasibility data to support a larger multi-ethnic randomized clinical trial on the effects of yoga on individuals with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-64; Pre- or Stage I hypertension with mean office blood pressure (two measurements using aneroid sphygmomanometer) of systolic between 120 and 159 mmHg or Diastolic between less than or equal to 80 and 99 [1]
* Medically stable on any current medications; BMI (kg/m2) between 18.5 - 40
* English speaking

Exclusion Criteria:

* Taking anti-hypertensive medication; Current use of insulin or oral hypoglycemic agents
* Previous cardiovascular event (prior myocardial infarction, stroke, or angina pectoris)
* Current or previous cancer diagnosis
* Congestive heart failure
* History of kidney disease
* Signs or symptoms of significant peripheral vascular disease
* Significant co-morbidities that preclude successful completion of the study
* Yoga practitioner (participated in more than 3 yoga sessions within the last year)

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure | Assessed within one week post a 12 week intervention
  24 hour ambulatory blood pressure: systolic, diastolic

SECONDARY OUTCOMES:
Psychosocial Stress | Assessed within one week after 12 week intervention
  perceived stress, coping, tolerance of uncertainty, sense of control,

CONTACTS AND LOCATIONS:
Overall Officials: Marshall A Hagins, PhD, PT, Principal Investigator — Long Island University
Locations (1):
- Long Island University, Brooklyn, New York, United States